CLINICAL TRIAL: NCT00823927
Title: Alveolar Macrophage Proteomics in HIV-associated Emphysema
Acronym: HIVE
Status: Completed | Type: Observational
Sponsor: Philip Diaz (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Philip Diaz, MD, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2005H0197; 2005H0197 (Other: The Ohio State University)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV; Emphysema; HIV Infections
Keywords: lung damage; cigarette smoking; HIV-seropositive; emphysema
MeSH Terms: conditions — Emphysema; HIV Infections; Cigarette Smoking; HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood lung fluid (optional)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Alveolar macrophage proteomes from HIV-seropositive smokers with emphysema
- 2: Alveolar macrophages proteomes of both HIV+ smokers without emphysema and HIV- smokers.

SUMMARY:
This study is being done to examine lung function changes in individuals with HIV infection and to understand why individuals with HIV have increased risk of lung damage from cigarette smoking.

DETAILED DESCRIPTION:
To delineate the natural history of HIV associated emphysema in the HAART era. To compare the alveolar macrophage proteomes from HIV-seropositive smokers with emphysema to the alveolar macrophages proteomes of both HIV+ smokers without emphysema and HIV- smokers.

To establish whether coinfection with HIV and Hepatitis C results in accelerated lung disease manifested by decrements in forced expiratory volume and carbon monoxide diffusing capacity.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable HIV-seropositive (and HIV-seronegative) individuals
* Ages 18 years and older
* Female subjects on no oral contraception with a negative pregnancy test
* Subjects capable of giving written consent

Exclusion Criteria:

* Known medical illness that would preclude bronchoscopy/BAL (e.g. unstable angina, new cardiac arrhythmia). This only pertains to subjects involved in the bronchoscopy phase of the study.
* Pregnant females
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2006-04-21 (Actual); Primary Completion 2008-06-23 (Actual); Study Completion 2008-06-23 (Actual)

PRIMARY OUTCOMES:
examine the natural history of smoking related lung damage in patients with HIV | 3 years
  HIV-Seropositive individuals are at increased risk of developing pulmonary emphysema (1,2). With improved therapy for HIV, and increased life expectancy in this population with a high smoking prevalence, chronic obstructive pulmonary disease (COPD) may assume an increasingly important role with respect to health related quality of life and medical complications. This research will provide a unique opportunity to examine the natural history of smoking related lung damage in patients with HIV infection. In addition, this research will involve sampling of lung cells to determine if there are unique proteins present that may be related to the increased risk of emphysema in this population. This may shed important insight into how the lung responds to injury and how it repairs itself. If critical proteins can be identified, treatment strategies may eventually be developed to either decrease proteins causing injury or increase protective proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Diaz, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States